CLINICAL TRIAL: NCT02797301
Title: A Computerised Test for Assessing the Early Reading Skills of Children With Mobility Limitations
Brief Title: A Computerised Test for Assessing the Early Reading Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Annie France Frère Slaets, PhD, University of Mogi das Cruzes
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 0135.0.237.000-10
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Learning Disorders
Keywords: early reading skills
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- synthetic test & computerised test (Experimental): Seventeen preschool children (G1), with no motor impairments, from a private school. The children in G1 performed the synthetic test before the computerised test.
  Interventions: Other: synthetic test; Other: computerised test
- computerised test & synthetic test (Experimental): Sixteen preschool children (G2), with no motor impairments, from a private school. The children in G2 performed the computerised test before the synthetic test.
  Interventions: Other: synthetic test; Other: computerised test
- computerised test (Experimental): Seven volunteers (G3), two males and five females, with moderate mobility impairment, patients from the Physical Therapy and Rehabilitation Clinic.
  Interventions: Other: computerised test

INTERVENTIONS:
Other: synthetic test — The children performed the synthetic test with no time restriction.
  Arms: computerised test & synthetic test; synthetic test & computerised test
Other: computerised test — The children performed the computerised test with no time restriction.

SUMMARY:
This study was to develop a computerised test with an adapted peripheral to assess the emerging literacy knowledge of children with mobility difficulties. The software was implemented using a game-like design controllable by a peripheral device without needing fine movements.

DETAILED DESCRIPTION:
Conventional tests for assessing the early reading skills of preschool children on school entry are not accessible to children with mobility limitations. This paper presents a game-like computerised test featuring an appealing scenario that is accessible to these children. It was developed on a platform that creates 2D vector graphics and contains three phases of interactive content accessible through an adapted peripheral. Conventional tests were also used to validate the effectiveness of the game. The two types of tests had the same degree of predictive power when completed by thirty three preschool children without mobility impairment.

ELIGIBILITY:
Inclusion Criteria:

* G1 and G2: preschool children; no motor difficulties and normal school performance.
* G3: with moderate mobility impairment; similar cognitive ages and notions of writing to the participants of groups G1 and G2; children between seven and seventeen years old.

Exclusion Criteria:

* G1 and G2: children who often miss classes; children between four and seven years.
* G3: no moderate mobility impairment

Ages: 4 Years to 17 Years | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Reading skills | 2 days
  The tests determine whether children can differentiate between the letters of the alphabet and squiggles, numbers, and mathematical signs (first phase); can realise that the same word can be written using uppercase, lowercase, and cursive letters (second phase); know the correct number of letters required to graphically represent the sounds used in speech (third phase). The numbers of incorrect choices made by children during the three phases of the computerised test (G1, G2 and G3) and the synthetic test (G1 and G2) are quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Annie F. Frère, PhD, Principal Investigator — University of Mogi das Cruzes

IPD SHARING:
Plan to Share IPD: No